CLINICAL TRIAL: NCT02582658
Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C -An Observational Study in Austria (REAL)
Brief Title: Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study in Austria (REAL)
Acronym: REAL
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-695
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2018-10

CONDITIONS: Chronic Hepatitis C
Keywords: Paritaprevir; Dasabuvir; Ombitasvir; Chronic Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic infection of HCV GT1 or GT4: Participants with confirmed chronic hepatitis C genotype (GT) 1 or 4, receiving combination therapy with the interferon-free ABBVIE REGIMEN (ombitasvir/paritaprevir/ritonavir +/- dasabuvir) ± Ribavirin (RBV) according to standard of care and in line with the current local label

SUMMARY:
The study seeks to provide evidence of the effectiveness and obtain patient reported outcome (PRO) and work productivity data of the interferon-free ABBVIE REGIMEN (ombitasvir/paritaprevir/ritonavir +/- dasabuvir) +/- Ribavirin (RBV) in chronic hepatitis C virus (HCV) infected participants in Austria.

ELIGIBILITY:
Inclusion Criteria:

Treatment-naïve or -experienced adult male or female patients with confirmed chronic hepatitis C, genotype (GT)1 or GT4, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± Ribavirin (RBV) according to standard of care and in line with the current local label

If RBV is co-administered with the ABBVIE REGIMEN, it has been prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy)

Patients must voluntarily sign and date a patient authorization to use and disclose his/her anonymized health data prior to inclusion into the study

Patient must not be participating or intending to participate in a concurrent interventional therapeutic trial

Exclusion Criteria:

none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic infection of HCV Genotype 1 (GT1) or Genotype 4 (GT4)
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2015-10-06; Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander P Dorr, PhD, Study Director — AbbVie Austria

REFERENCES:
- [Derived] Ferenci P, Bourgeois S, Buggisch P, Norris S, Curescu M, Larrey D, Marra F, Kleine H, Dorr P, Charafeddine M, Crown E, Bondin M, Back D, Flisiak R. Real-world safety and effectiveness of ombitasvir/paritaprevir/ritonavir +/- dasabuvir +/- ribavirin in hepatitis C virus genotype 1- and 4-infected patients with diverse comorbidities and comedications: A pooled analysis of post-marketing observational studies from 13 countries. J Viral Hepat. 2019 Jun;26(6):685-696. doi: 10.1111/jvh.13080. Epub 2019 Mar 5. PMID 30739368
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 173 patients were enrolled in the study; 2 patients never started treatment and were excluded from the safety (SP; N=171); 6 patients were excluded from the core population (CP; N=165), defined as all SP patients who met eligibility criteria and were adequately treated according to the standard of care and local label recommendations.
Groups:
- ABBVIE REGIMEN +/- Ribavirin (RBV): ABBVIE REGIMEN ± Ribavirin (RBV) according to standard of care and in line with the current local label where ABBVIE REGIMEN included ombitasvir/paritaprevir/ritonavir +/- dasabuvir
Period: Overall Study
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Started | 171
Completed | 146
Not Completed | 25
Not completed — Failure to Return | 10
Not completed — Insufficient Virological Response | 2
Not completed — Withdrawn Consent | 1
Not completed — Death | 1
Not completed — Not further specified | 11

BASELINE CHARACTERISTICS:
Population: The Core Population (CP) was defined as all patients in the safety population (SP; all enrolled subjects who received at least 1 dose of study drug) who met eligibility criteria and were adequately treated according to the standard of care and within local label recommendations.
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasin | 158
  Asian/Oriental | 4
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) levels < 50 IU/mL 12 weeks after the last actual dose of study drug.
Time Frame: 12 Weeks after the last dose of study drug
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
percentage of participants | 84.8 [78.6 to 89.5]

2. Secondary Outcome: Percentage of Participants With Virological Response at End of Treatment (EoTR)
Description: The percentage of participants with virological response (HCV RNA <50 IU/mL) at end of treatment (EoT, defined as last intake of ABBVIE REGIMEN or ribavirin [RBV]).
Time Frame: Up to 24 weeks of treatment
Population: Core Population (CP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
percentage of participants | 94.5 [90.0 to 97.1]

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure (Breakthrough)
Description: The percentage of participants with on-treatment virologic failure (breakthrough [defined as at least one documented HCV RNA <50 IU/mL followed by HCV RNA >= 50 IU/mL during treatment]).
Time Frame: Up to approximately 24 weeks
Population: Core Population (CP)
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
percentage of participants | 1.2

4. Secondary Outcome: Percentage of Participants Achieving SVR12 (Core Population Sufficient Follow-up)
Description: SVR12 is defined as HCV RNA levels < 50 IU/mL 12 weeks after the last actual dose of study drug in the Core Population Sufficient Follow-up (CPSFU).
Time Frame: 12 weeks after last dose of study drug
Population: CP subjects with evaluable HCV RNA data ≥70 days after last dose AbbVie Regimen, or HCV RNA value ≥50IU/mL at last measurement postbaseline, or HCV RNA <50IU /mL at last measurement postbaseline, but no HCV RNA value ≥70 days after last dose AbbVie Regimen due to safety or virologic failure (relapse reported but date/value of HCV RNA test missing).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 146
percentage of participants | 95.9 [91.3 to 98.1]

5. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: The percentage of participants with relapse (defined as HCV RNA <50 IU/mL at EoT followed by HCV RNA ≥50 IU/mL)
Time Frame: Up to 12 weeks after last dose of study drug
Population: Core Population (CP)
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
percentage of participants | 0.0

6. Other Pre Specified Outcome: Percentage of Planned Duration of Ribavirin (RBV) Taken
Description: Adherence to RBV is defined as percentage of target dose (adherence=cumulated dose taken/ [initially prescribed dose x planned duration]).
Time Frame: Up to 24 weeks of treatment
Population: All participants in the Core Population (CP) who received RBV
Measure: Mean (Standard Deviation); unit: percentage of planned RBV dose taken
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 60
percentage of planned RBV dose taken | 95.7 (16.96)

7. Other Pre Specified Outcome: Total Score of Participant Activation According to the Patient Activation Measure (PAM-13) Questionnaire
Description: The PAM-13 item scale is a measure used to assess the patient knowledge, skill, and confidence for self-management. Each of the 13 items can be answered with one of four possible response options, which are "disagree strongly" (1), "disagree" (2), "agree" (3), "agree strongly" (4). Responses are summed and averaged to come up with an overall score of level 1 through level 4. The responses to the 13 questions are summed and transformed into a PAM Score between 0 and 100; a higher score indicates more knowledge and confidence to take action for self-management.
Time Frame: Day 0 and End of Treatment (EoT)
Population: Core Population (CP)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
score on a scale
  PAM-13 Day 0: number analyzed (Participants) | 122
  PAM-13 Day 0 | 63.3 (10.9)
  PAM-13 EOT: number analyzed (Participants) | 77
  PAM-13 EOT | 62.6 (10.3)

8. Other Pre Specified Outcome: Percentage of Participants With Concomitant Medications
Description: Percentage of participants taking at least 1 concomitant medication
Time Frame: Day 0 to end of treatment (up to 24 weeks)
Population: The safety population (SP) was defined as enrolled patients who received at least 1 dose of ABBVIE REGIMEN.
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 171
percentage of participants
  Patients Taking at least 1 co-medication | 49.1
  Analgesics | 12.3
  Antidepressants | 11.7
  Beta blocking agents | 9.9
  Calcium channel blockers | 8.8
  Thyroid therapy | 7.6
  Vitamins | 5.8
  Blood glucose lowering drugs | 4.7
  Drugs used in addictive disorders | 4.7
  ACE inhibitors | 4.1
  Angriotensin II antagonists | 4.1
  Anti-asthmatics | 4.1
  Benzodiazepine derivatives | 4.1
  Antithrombotic | 3.5
  Drugs for peptic ulcer/gastroesophageal reflux dis | 3.5
  Angiotensin II Antagonists | 2.9
  Antipsychotics | 2.9
  Diuretics | 2.9
  ACE inhibitors, combinations | 2.3
  Insulin and analogues | 2.3
  Mineral supplements | 2.3
  Antieplieptics | 1.8
  Anti-inflammatory and antirheumatic products | 1.8
  Drugs used in benign prostatic hypertrophy | 1.8
  Herbal medicine | 1.8
  Vasodilators for cardiac diseases | 1.8
  Anti-dementia drugs | 1.2
  Antibacterials | 1.2
  Anti-gout preparations | 1.2
  Drugs for functional gastrointestinal disorders | 1.2
  HMG COA reductase inhibitors | 1.2
  Hypnotics and sedatives | 1.2
  Immunosuppressive agents | 1.2
  Lipotropics | 1.2
  Vasoprotectives | 1.2
  Anti-adrenergic antihypertensives | 0.6
  Antibiotics for dermatological use | 0.6
  Antiemetics and anti nauseants | 0.6
  Antigloucoma | 0.6
  Antihistamines | 0.6
  Antineoplastic/immunomodulating agents, cytostatic | 0.6

9. Other Pre Specified Outcome: Percentage of Participants With Co-morbidities and/or Co-infections
Description: Percentage of participants with co-morbidities and/or co-infections at baseline (Day 0).
Time Frame: Day 0
Population: Core Population (CP)
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
percentage of participants
  All co-morbidities and co-infections | 57.6
  HCV co-infections | 1.8
  Liver and/or CHC related co-morbidities | 5.5
  Chronic kidney disease | 3.0
  Psychiatric disorders | 15.2
  Diabetes mellitus | 9.7
  Lipid disorder | 5.5
  Hyperthyroidism | 0.6
  Hypothyroidism | 8.5
  Cardiovascular disease | 23.0
  Immunologically medicated disease | 1.2
  Psychoactive substance dependency | 10.9
  Other | 20.6

10. Other Pre Specified Outcome: Quality of Life Measured With the EuroQol 5 Dimension 5 Level (EQ-5D-5L) Questionnaire
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status (utility). The 5 items in the EQ-5D-5L comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) to describe the subject's current health state. Each dimension comprises 5 levels with corresponding numeric scores, where 1 indicates no problems, and 5 indicates extreme problems. A unique EQ-5D-5L health state is defined by combining the numeric level scores for each of the 5 dimensions and the total score is normalized from -0.594 to 1.000, with higher scores representing a better health state. An increase in the EQ-5D-5L total score indicates improvement. The EQ-5D visual analogue scale (VAS) records the participant's self-rated health status on a vertical graduated scale from 0 to 100, with 0 indicating the worst imaginable health state and 100 indicating the best imaginable health state. An increase in EQ-5D-5L VAS score indicates improvement.
Time Frame: Day 0 and post treatment week 12
Population: Core Population (CP)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
score on a scale
  EQ-5D-5L: Index Score Basline: number analyzed (Participants) | 142
  EQ-5D-5L: Index Score Basline | 0.83 (0.17)
  EQ-5D-5L: Index Score 12 Weeks EOT: number analyzed (Participants) | 99
  EQ-5D-5L: Index Score 12 Weeks EOT | 0.88 (0.15)
  EQ-5D-5L: VAS Score Basline: number analyzed (Participants) | 151
  EQ-5D-5L: VAS Score Basline | 70.4 (19.5)
  EQ-5D-5L: VAS Score 12 Weeks EOT: number analyzed (Participants) | 106
  EQ-5D-5L: VAS Score 12 Weeks EOT | 79.4 (17.3)

11. Other Pre Specified Outcome: Change in Mean Score From Baseline to 12 Weeks After End of Treatment (EOT) in Work Productivity and Activity Impairment (WPAI) Version 2: Hepatitis C Questionnaire
Description: The WPAI questionnaire was used to measure work absenteeism, work presenteeism, work productivity impairment and daily activity impairment. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity: Presenteeism - percentage of impairment while working due to health problem; Total work productivity impairment - percentage of overall work impairment due to health problem Absenteeism - percentage of work time missed due to health problem; Total activity impairment - percentage of general (non-work) activity impairment due to health problem
Time Frame: Day 0 to post treatment week 12
Population: Core Population (CP)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
percentage
  Change from baseline in absenteeism: number analyzed (Participants) | 32
  Change from baseline in absenteeism | 0.1 (0.4)
  Change from baseline in presenteeism: number analyzed (Participants) | 31
  Change from baseline in presenteeism | -10.6 (17.3)
  Change from baseline in total work impairment: number analyzed (Participants) | 31
  Change from baseline in total work impairment | -10.5 (17.2)
  Change from baseline in total activity impairment: number analyzed (Participants) | 83
  Change from baseline in total activity impairment | -8.3 (29.5)

12. Other Pre Specified Outcome: Patient Support Program (PSP) Utilization and Satisfaction Assessment
Description: The AbbVie PSP included educational and information material (including printed, online, pillbox), digital and mobile resource (web-portal), digital and mobile resources (reminders). The PSP utilization and satisfaction assessment evaluated the frequency of utilization (usually daily, several times per week, usually once weekly, less than once weekly) and patient's overall satisfaction (very good, good, satisfactory) with their respective PSP.
Time Frame: Up to 24 weeks of treatment
Population: Core Population (CP)
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 26
percentage of participants
  Participants Using at least 1 PSP since last visit | 65.4
  Personal support - satisfaction Very Good | 34.6
  Personal support satisfaction - Good | 7.7
  Personal support satisfaction - Satisfactory | 3.8

13. Other Pre Specified Outcome: Percentage of Participants With Adherence to Planned RBV Target Dose Taken
Description: Adherence to RBV is defined as percentage of target dose (adherence=cumulated number of pills taken / [initially prescribed number of pills x planned duration]) and categorized as follows: >105%, >95% - <=105%, >80% - <=95%, >50% - <=80%, <=50%.
Time Frame: Up to 24 weeks of treatment
Population: All participants in the Core Population (CP) who received RBV
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 60
percentage of participants
  > 105% Adherence | 3.3
  >95% - <=105% Adherence | 85.0
  >80% - <=95% Adherence | 1.7
  >50% - <=80% Adherence | 5.0
  <=50% Adherence | 5.0

14. Other Pre Specified Outcome: Percentage of Participants Deviating From the Target ABBVIE Regimen Duration
Description: Deviations from the target dose of the ABBVIE REGIMEN were defined as the actual duration is shortened/prolonged (exceedence) for more than 7 days.
Time Frame: Up to 24 weeks of treatment
Population: Core Population (CP)
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
percentage of participants
  Early discontinuation | 7.9
  Exeedance | 1.8
  Not deviated | 90.3

15. Other Pre Specified Outcome: Percentage of Participants With Adherence to Planned ABBVIE Regimen Target Dose Taken
Description: Adherence to the ABBVIE REGIMEN was defined as percentage of target dose (adherence=cumulated number of pills taken / [initially prescribed number of pills x planned duration]) and categorized as follows: >105%, >95% to <=105%, >80% to <=95%, >50% to <=80%, <=50%.
Time Frame: Up to 24 weeks of treatment
Population: Core Population (CP)
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Number analyzed (Participants) | 165
percentage of participants
  > 105% Adherence | 1.8
  >95% - <=105% Adherence | 88.5
  >80% - <=95% Adherence | 3.0
  >50% - <=80% Adherence | 3.6
  <=50% Adherence | 3.0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 30 days post-study drug dosing (up to 28 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug.
Arm/Group | ABBVIE REGIMEN +/- Ribavirin (RBV)
Serious Adverse Events (participants affected / at risk) | 5/171
Other Adverse Events (participants affected / at risk) | 27/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABBVIE REGIMEN +/- Ribavirin (RBV) (N=171)
Diarrhea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Fatigue (General disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABBVIE REGIMEN +/- Ribavirin (RBV) (N=171)
Fatigue (General disorders) | 13
Nausea (Gastrointestinal disorders) | 7
Headache (Nervous system disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.